CLINICAL TRIAL: NCT00113126
Title: A Randomized Trial of CD4 Guided Treatment Interruption, Compared to Continuous Treatment, for HIV Infection
Brief Title: Staccato: A Trial of CD4 Guided Treatment Interruption, Compared to Continuous Treatment, for HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCS # 356
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2005-06

CONDITIONS: HIV Infection; AIDS
Keywords: Scheduled treatment interruptions; STI
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Treatment Interruption

INTERVENTIONS:
Drug: Treatment interruption

SUMMARY:
Treatment of HIV repairs the immune system, but continuous treatment is expensive and causes side effects. Would it not be better to treat intermittently, e.g. stop treatment when the immune system has recovered, and start again only when damage reappears? That is the question which STACCATO proposes to answer.

Approximately 500 patients were recruited for this trial from 2002 to 2004. One third were treated continuously; in two thirds, the treatment was interrupted whenever the CD4 count, a measure of immune recovery, exceeded 350. At the end of 2005, the two treatment groups will be compared in order to see which fared better regarding amount of drugs used, side effects, CD4 counts, and development of resistance to treatment.

DETAILED DESCRIPTION:
Continuous treatment has been very successful in diminishing the diseases and deaths caused by HIV. However, continuous treatment is expensive. Intermittent treatment will always cost less than continuous treatment, and therefore has the potential to facilitate access to highly active antiretroviral therapy (HAART) in developing countries. HAART also causes many undesirable effects. Intermittent treatment decreases exposure to drugs and is therefore expected to decrease side effects.

STACCATO is a randomised trial of intermittent versus continuous anti-retroviral treatment. At least 600 patients on HAART, with viremia below 50 copies/ml and CD4 count above 350 cells/ml were randomised to one of two arms, in 1:2 proportions:

* Arm 1: Continuation (control) arm: Drugs are continued or changed according to current guidelines and good clinical practice.
* Arm 2: CD4-guided arm: Drugs discontinued and reintroduced according to CD4 counts, with HAART being administered only if CD4 count is < 350 cells/ml.

Randomized treatment will continue during an average of approximately 2 years, and will be followed by a period of 12 to 24 weeks' continuous treatment, for patients in both arms.

Endpoints: The amount of drugs used, side effects, viremia and CD4 counts, number of clinical events, at the end of the randomized treatment period, and again 12 to 24 weeks later. A subproject will study the effect of treatment interruption on resistance development, mutations in proviral DNA and proviral DNA levels.

ELIGIBILITY:
Inclusion Criteria:

* CD4 lymphocyte count above 350/microliter and viral HIV1-RNA below 50 copies/ml on antiretroviral treatment.

Exclusion Criteria:

* Virologic failure of treatment. Failure of treatment defined as a treatment switch motivated by high viral loads on treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526
Dates: Start 2002-01; Study Completion 2005-10

PRIMARY OUTCOMES:
Amounts of drugs used
Response of viral load to retreatment after interruption

SECONDARY OUTCOMES:
Opportunistic infections and deaths
Adverse effects
CD4 counts
Resistance development

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Hirschel, MD, Study Chair — Infectious Diseases Unit - University Hospital
Locations (1):
- Infectious Diseases Unit - University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Ananworanich J, Nuesch R, Le Braz M, Chetchotisakd P, Vibhagool A, Wicharuk S, Ruxrungtham K, Furrer H, Cooper D, Hirschel B, Bernasconi E, Cavassini M, Ebnother C, Fagard C, Genne D, Khanna N, Perrin L, Phanupak P, Ubolyam S, Vernazza P, Yerly S; Swiss HIV Cohort Study. Failures of 1 week on, 1 week off antiretroviral therapies in a randomized trial. AIDS. 2003 Oct 17;17(15):F33-7. doi: 10.1097/00002030-200310170-00001. PMID 14523294
- [Result] Ananworanich J, Gayet-Ageron A, Le Braz M, Prasithsirikul W, Chetchotisakd P, Kiertiburanakul S, Munsakul W, Raksakulkarn P, Tansuphasawasdikul S, Sirivichayakul S, Cavassini M, Karrer U, Genne D, Nuesch R, Vernazza P, Bernasconi E, Leduc D, Satchell C, Yerly S, Perrin L, Hill A, Perneger T, Phanuphak P, Furrer H, Cooper D, Ruxrungtham K, Hirschel B; Staccato Study Group; Swiss HIV Cohort Study. CD4-guided scheduled treatment interruptions compared with continuous therapy for patients infected with HIV-1: results of the Staccato randomised trial. Lancet. 2006 Aug 5;368(9534):459-65. doi: 10.1016/S0140-6736(06)69153-8. PMID 16890832
- [Derived] Calmy A, Gayet-Ageron A, Montecucco F, Nguyen A, Mach F, Burger F, Ubolyam S, Carr A, Ruxungtham K, Hirschel B, Ananworanich J; STACCATO Study Group. HIV increases markers of cardiovascular risk: results from a randomized, treatment interruption trial. AIDS. 2009 May 15;23(8):929-39. doi: 10.1097/qad.0b013e32832995fa. PMID 19425222
- [Derived] Ananworanich J, Nuesch R, Cote HC, Kerr SJ, Hill A, Jupimai T, Laopraynak N, Saenawat S, Ruxrungtham K, Hirschel B. Changes in metabolic toxicity after switching from stavudine/didanosine to tenofovir/lamivudine--a Staccato trial substudy. J Antimicrob Chemother. 2008 Jun;61(6):1340-3. doi: 10.1093/jac/dkn097. Epub 2008 Mar 12. PMID 18339636